CLINICAL TRIAL: NCT00646061
Title: Pain Control in Renal Colic
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Seoul National University Hospital, Seoul National University Hospital
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: B-0705/045-005
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Last update posted 2009-09-22 (Estimated); Status verified 2009-09

CONDITIONS: Renal Colic
Keywords: renal colic
MeSH Terms: conditions — Renal Colic | interventions — Butylscopolammonium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): morphine, ketorolac, and buscopan
  Interventions: Drug: buscopan
- 2 (No Intervention): morphine and ketorolac

INTERVENTIONS:
Drug: buscopan
  Arms: 1

SUMMARY:
Renal colic is very common in emergency department patients. Our aim of this study is which combination of drug is more effective in renal colic.

ELIGIBILITY:
Inclusion Criteria:

* adult, clinical suspicion of renal colic

Exclusion Criteria:

* under 15
* do not consent
* contraindication of morphine, ketorolac, or buscopan
* previously pain controlled

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2007-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
pain control

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Kyeongi-do, South Korea